CLINICAL TRIAL: NCT02800551
Title: Dose-intensified Image-guided Fractionated Stereotactic Body Radiation Therapy for Painful Spinal Metastases Versus Conventional Radiation Therapy: a Randomised Controlled Trial (DOSIS RCT)
Brief Title: Clinical Trial Comparing Dose-intensified SBRT With Conventional Radiation Therapy for Spinal Metastases
Acronym: DOSIS RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOSIS RCT
Record Dates: First submitted 2016-04-29; First posted 2016-06-15 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Spinal Metastasis
MeSH Terms: interventions — Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SBRT (Arm A) (Experimental): dose-intensified image-guided SBRT using simultaneous integrated boost:
  * in the case of no epidural involvement: 40 Gy and 20 Gy in 5 fractions to the high-dose and conventional-dose target volume, respectively.
  * In the case epidural involvement: 48.5 Gy and 30 Gy in 10 fractions to the high-dose and conventional-dose target volume, respectively.
  Interventions: Radiation: dose-intensified image-guided SBRT using simultaneous integrated boost
- Conventional Radiation Therapy (Arm B) (Active Comparator): External 3-dimensional conformal radiotherapy (3D-CRT):
  Homogeneous irradiation of the affected vertebra delivering either
  * 20 Gy in 5 fractions or
  * 30 Gy in 10 fractions.
  Interventions: Radiation: External 3-dimensional conformal radiotherapy (3D-CRT)
- SBRT (prospective observational) (Experimental): Patients eligible for the prospective observational arm will be treated according to the investigational arm (arm A) of the randomised arm of the trial.
  Interventions: Radiation: dose-intensified image-guided SBRT using simultaneous integrated boost

INTERVENTIONS:
Radiation: dose-intensified image-guided SBRT using simultaneous integrated boost
  Arms: SBRT (Arm A); SBRT (prospective observational)
Radiation: External 3-dimensional conformal radiotherapy (3D-CRT)
  Arms: Conventional Radiation Therapy (Arm B)

SUMMARY:
This study will compare pain (primary end-point) and local metastatic tumor control (secondary end-point) after dose-intensified image-guided fractionated stereotactic body radiation therapy (SBRT) for painful mass-type spinal metastases versus conventional radiation therapy.

DETAILED DESCRIPTION:
Rationale: Radiation therapy is an effective palliative treatment for painful spinal metastases. A sub-group of patients with mass-type spinal metastases, a factor associated with poor local metastasis control, require treatment optimization ensuring durable pain control and metastatic tumor control.

Proposed solution: To intensify (escalate) radiation dose using simultaneous integrated boost with image-guided hypofractionated SBRT for painful mass-type spinal metastases in a randomized controlled trial. Two experimental fractionation regimes will be tested in the study depending on presence or absence of epidural involvement. Dose intensification is expected to achieve long-term pain control and long-term palliation as well as long-term local metastatic tumor control without adding toxicity as compared to conventional fractionation regimes with conventional radiation therapy.

The study will be carried out as multinational, multicentre phase II clinical controlled trial enrolling patients with painful mass-type spinal metastases who are eligible for radiation therapy without surgery. This study additionally includes a prospective observational arm for patients not eligible for randomisation who are treated in analogy to arm A of the randomised arm.

ELIGIBILITY:
Inclusion Criteria:

* Established histological diagnosis of a malignant primary or metastatic tumor;
* Histologically, radiologically or scintigraphically proven spinal metastasis;
* Pain in the affected spinal region or free of pain under pain medication;
* Age ≥18 years old;
* Karnofsky performance status ≥60%;
* Written informed consent.

Exclusion Criteria:

* Modified Bauer Score < 2;
* No-mass-type metastatic lesion, defined as a 3D space-occupying lesion visible on CT and/or MR;
* "Radiosensitive" histology of the primary tumor, e.g., lymphoma, small-cell lung cancer, multiple myeloma, germ cell tumors;
* Progressive neurological symptoms/deficit;
* More than 3 affected vertebrae in one target site;
* More than 2 treatment sites;
* Spinal Instability Neoplastic Score (SINS) 13 - 18, i.e., unstable;
* Unable to tolerate treatment (unable to lie flat and immobilized);
* Previous radiotherapy of the region at the level of the affected vertebrae;
* Previous radionuclide therapy within 30 days before stereotactic body radiation therapy;
* Previous surgery (stabilization) of the affected vertebrae;
* Contraindications for MR scanning, e.g., pacemakers;
* Patients with allergy to contrast agents used in computer tomography (CT) and magnetic resonance (MR) imaging or patients who cannot be premedicated to use contrast agent;
* Pregnant or lactating women;
* Women of child bearing potential or sexually active males not willing to use effective contraception while on treatment and 3 months after the end of treatment;
* Mental conditions rendering the patient unable to understand the nature, scope, and possible consequences of the study;
* Patient unlikely to comply with protocol, i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Pain response - improvement by ≥ 2 points on the pain Visual Analogue Scale at 6 months post-treatment at the treatment site | 6 months

SECONDARY OUTCOMES:
Local metastasis control | up to 2 years
  Local metastasis control is defined from the day of randomization to a day of local (at the site of the treated spinal metastasis) progression, i.e. local failure, determined on control MR images as a change in signal intensity or on CT images as increasing soft-tissue mass. Increased epidural disease or enlargement of paraspinal disease on control images will be documented as progression.
Overall survival | up to 2 years
  Overall survival is defined from the day of randomization to a day of death of any cause.
Cancer-specific survival | up to 2 years
  Cancer-specific survival is defined from the day of randomization to a day of death due to cancer progression.
Quality-of-life (QoL) | Day 1 and last day of treatment (usually day5 if Radiotherapy is delivered in 5 fractions, and day 12 if Radiotherapy is delivered in 10 fractions); months 1, 3, 6, 9, 12, 18 and 24
  Quality-of-life (QoL) as measured by the EORTC QLQ-C15-PL, EORTC-BM22 and EQ-5D-5L patient reported questionnaires
Epidural spinal cord compression | up to 2 years
  Epidural spinal cord compression (ESCC) will be scored using Bilsky criteria.
Acute and late toxicity | Acute toxicity: up to 3 months; late toxicity: from 3 months up to 24 months
  Acute aund late toxicity will be assessed in accordance to NCI CTCEA version 4.03 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, Prof. Dr., Principal Investigator — Universitätsspital Zürich
Locations (1):
- UniversitätsSpital Zürich, Klinik für Radio-Onkologie, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No